CLINICAL TRIAL: NCT01436032
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Analgesic Efficacy, Safety and Tolerability of Intravenous N1539 in Subjects After Abdominal Laparoscopic Surgery
Brief Title: Efficacy, Safety and Tolerability Study of N1539 in Subjects After Abdominal Laparoscopic Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N1539-05
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Laparoscopic Surgery
MeSH Terms: interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- N1539 15 mg (Experimental)
  Interventions: Drug: N1539
- N1539 30 mg (Experimental)
  Interventions: Drug: N1539
- Ketorolac (Active Comparator): IV
  Interventions: Drug: Ketorolac Tromethamine
- Placebo (Placebo Comparator): IV
  Interventions: Drug: Placebo
- N1539 7.5mg (Experimental)
  Interventions: Drug: N1539

INTERVENTIONS:
Drug: N1539 — IV
  Arms: N1539 7.5mg
Drug: N1539 — IV
  Arms: N1539 15 mg
Drug: N1539 — IV
  Arms: N1539 30 mg
Drug: Ketorolac Tromethamine — IV
  Arms: Ketorolac
Drug: Placebo — IV
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the analgesic efficacy and safety of N1539 in subjects undergoing abdominal laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo elective abdominal laparoscopic surgery involving a single site/organ and does not have intraperitoneal metastases suspected or identified

Exclusion Criteria:

* Use of ketorolac is contraindicated
* Use of general anesthesia is contraindicated
* Has a medical condition that could adversely impact subject participation
* Has diabetes mellitus and glycosylated hemoglobin (HbA1c) >9.5 or history of prolonged uncontrolled diabetes
* Body mass index (BMI) less than 18 or greater than 35
* Has a history of intolerance or allergic reactions to non-steroidal anti-inflammatory drugs (NSAIDs), Cox-2 inhibitors, aspirin or other salicylates
* Known or suspected sleep apnea
* History of Hepatitis B or C
* Has a psychiatric disorder that impairs capability of subject to report pain
* Known to have chronic obstructive pulmonary disease (COPD) with carbon dioxide retention or chronic hypoxemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Sum of the time-weighted pain intensity differences (SPID) as recorded on the Visual Analog Scale (VAS) from baseline (time 0) to 24 hours following the first dose of study medication (SPID 24) | 0 to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (1):
- Lotus Clinical Research LLC, Pasadena, California, United States

REFERENCES:
- [Derived] Viscusi ER, Gan TJ, Bergese S, Singla N, Mack RJ, McCallum SW, Du W, Hobson S. Intravenous meloxicam for the treatment of moderate to severe acute pain: a pooled analysis of safety and opioid-reducing effects. Reg Anesth Pain Med. 2019 Mar;44(3):360-368. doi: 10.1136/rapm-2018-100184. Epub 2019 Feb 7. PMID 30737315